CLINICAL TRIAL: NCT05066698
Title: A Phase 2b, Multi-Center, Randomized, Double-Blind, Placebo-Controlled Study With Open-Label Extension to Evaluate the Safety and Efficacy of ST266 Eye Drops in the Treatment of Persistent Corneal Epithelial Defects
Brief Title: ST266 Eyedrops for the Treatment of Persistent Corneal Epithelial Defects
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor undergoing financial hardships - no longer able to support trial; no safety concerns.
Sponsor: Noveome Biotherapeutics, formerly Stemnion (Industry)
Collaborators: IQVIA Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ST266-PED-202
Record Dates: First submitted 2021-09-23; First posted 2021-10-04 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Persistent Corneal Epithelial Defect

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blind, Placebo-Controlled trial with Open-Label Extension
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ST266 (Experimental): Topical ocular application: one drop in the study eye four times a day for 8 weeks
  Interventions: Biological: ST266; Biological: Open-label ST266
- Placebo (Placebo Comparator): Topical ocular application: one drop in the study eye four times a day for 8 weeks
  Interventions: Other: 0.67% Sodium Chloride Ophthalmic Solution; Biological: Open-label ST266

INTERVENTIONS:
Biological: ST266 — Topical ocular application: one drop four times a day for eight weeks
  Arms: ST266
Other: 0.67% Sodium Chloride Ophthalmic Solution — Topical ocular application: one drop four times a day for eight weeks
  Other Names: Placebo
  Arms: Placebo
Biological: Open-label ST266 — Open label extension for non-healers after completion of double-blind treatment phase: topical ocular application of one drop four times a day for eight weeks

SUMMARY:
The primary objective is to determine the efficacy of ST266 eye drops in healing persistent epithelial defects (PED). After 8 weeks of randomized, double-blind treatment, non-healers will enter into an additional 8-week open-label ST266 treatment period. All patients will be followed for 3-months post-treatment for monitoring of safety and maintenance of re-epithelialization.

ELIGIBILITY:
Inclusion Criteria:

1. Male and non-pregnant/non-breastfeeding female subjects aged 18 years and older.
2. Subjects with a PED present for at least seven (7) days at the time of Screening.
3. The defect must be at least 1.0 mm (longest linear measurement) at Screening and Baseline (Day 1) and must be measurable by slit lamp.
4. In the Investigator's opinion, the defect is persistent i.e., the defect has not shown improvement despite conventional treatment such as tear supplements and bandage contact lenses.
5. The original defect to the cornea must be the result of an injury, infection, disease, or surgery to the eye.

Exclusion Criteria:

1. Diabetic cohort only: enrollment will be limited to include up to 50% of subjects with diabetes, as indicated by HbA1c level >6.5%. Subjects with a HbA1c level >6.5% after closure of the diabetic cohort will be excluded.
2. Subjects currently being treated with cenegermin or other rhNGF in the study eye.
3. Subjects currently using topical antibiotic eye drops in the study eye. Subjects on current antibiotic therapy must be willing to switch to study-provided moxifloxacin.
4. Subjects currently taking topical steroids or corticosteroid-containing eye drops or ointment in the study eye. Subjects currently taking systemic corticosteroids with a dose of >10mg/day prednisone or equivalent.
5. Subjects currently using topical antihistamine eye drops or vasoconstrictors in the study eye.
6. Subjects currently using topical or local immunosuppressive agents (e.g., optic cyclosporine or lifitegrast) in the study eye.
7. Subjects who require treatment with autologous serum eyedrops or amnion products in the study eye.
8. Subjects who need to use contact lenses for refractive correction during the study.
9. Subjects who require treatment with bandage contact lens or punctal plugs in the study eye that cannot be removed.
10. Subjects currently taking antiviral medications for an active infection in the study eye. Subjects taking antiviral medications for prophylaxis may be enrolled in the study at the Investigator's discretion, provided that the subject remain on a stable dosing regimen throughout the duration of the study.
11. History of ocular surgery (including laser or refractive surgery) in the study eye within 1 month prior to study screening or, in the opinion of the Investigator, there are persistent post-surgical complications that would impact the study data.
12. Subjects with an uncontrolled lid or ocular infection in the study eye.
13. History of alkali burns of the cornea.
14. The circumference affected by limbal blood vessel ischemia is greater than 75 percent of the limbal circulation.
15. Subjects with severe lid abnormalities contributory to the persistence of the PED such as inability to close the lids.
16. Subjects who have a history of AIDS or HIV.
17. Subjects who have participated in a clinical trial (including a previous study involving ST266) within 30 days prior to Day 1.
18. Subjects who have more than one distinct PED in the study eye prior to screening visits. Subjects who develop PEDs after the screening visit will remain in the study; however, only the original study PED will be assessed.
19. For subjects with bilateral PEDs, only the eye with the larger PED should be entered into the study. The non-study eye will receive standard of care treatment and be observed throughout the trial.
20. Subjects with bullous keratopathy in the study eye.
21. Subjects with corneal perforation or impending corneal perforation in the study eye.
22. Subjects with uncontrolled glaucoma.
23. Female subjects who are pregnant or breastfeeding. Female subjects who are neither postmenopausal for at least 1 year nor surgically sterile require a negative urine pregnancy test. All subjects must use an acceptable form of birth control during the study such as abstinence, barrier method, or hormonal contraceptive.
24. Epithelial defect was classified as a progressive corneal melt caused by an immunological process such as rheumatoid melt or Mooren's ulceration.
25. Subjects with recurrent corneal erosion or corneal basement membrane dystrophy.
26. Known hypersensitivity to study provided lubricating drops, antibiotic drops, and/or procedural medications such as fluorescein dye.
27. Consideration by the Investigator, for any reason, that the subject is an unsuitable candidate to receive ST266.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-04-27 (Actual); Primary Completion 2022-09-07 (Actual); Study Completion 2022-09-07 (Actual)

PRIMARY OUTCOMES:
Clinical Success | 8 weeks
  Proportion of subjects with clinical success between ST266 and placebo arms, defined as complete re-epithelialization of the corneal epithelial defect by week 8 of treatment.

SECONDARY OUTCOMES:
Safety of ST266 | 7 months
  Incidence of Adverse Events (AEs) and Serious Adverse Events (SAEs) in subjects treated with ST266 versus placebo
Time to re-epithelialization | 8 weeks
  Time (in days) to first complete re-epithelization of PED in subjects treated with ST266 versus placebo.
Maintenance of re-epithelialization during treatment | 8 weeks
  Time (in days) of re-epithelialization maintenance during treatment.
Maintenance of re-epithelialization post-treatment | 12 weeks
  Maintenance of corneal re-epithelization at 2 weeks and up to 12 weeks after the end of treatment in subjects treated with ST266 versus placebo.
Change in BCVA from Baseline | 7 months
  Mean change in Best Corrected Visual Acuity (BCVA) from Baseline over time and maintenance up to 12 weeks after the end of treatment in subjects treated with ST266 versus placebo.
Incidence of Rescue Therapy | 8 weeks
  Incidence of need for rescue within 8 weeks in subjects treated with ST266 versus placebo.
Clinical Success in Open-Label Extension | 8 weeks
  Proportion of subjects with complete re-epithelization of the corneal epithelial defect after 8 weeks of open label treatment based on the Independent Reading Center (IRC) image assessment.
Use of Lubricating Drops | 8 weeks
  Mean usage of preservative-free lubricating drops used for comfort in subjects treated with ST266 versus placebo.
VAS Score | 8 weeks
  Mean change in Visual Analog Scale (VAS) score from Baseline over time in subjects treated with ST266 versus placebo.
Size of Defect | 7 months
  Size of epithelial defect

CONTACTS AND LOCATIONS:
Locations (31):
- United States (31):
  - Trinity Research Group, Dothan, Alabama
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Atlantis Eye Care, Huntington Beach, California
  - UCLA Stein Eye Institute, Los Angeles, California
  - Stanford, Palo Alto, California
  - UCLA Doheny Eye Center, Pasadena, California
  - California Eye Specialists Medical Group, Pasadena, California
  - Bowden Eye & Associates, Jacksonville, Florida
  - Shettle Eye Research, Largo, Florida
  - Millennium Clinical Research, Inc, Miami, Florida
  - MedEye Associates, Miami, Florida
  - Cincinnati Eye Institute, Edgewood, Kentucky
  - University of Maryland Eye Associates, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts Eye and Ear, Boston, Massachusetts
  - Mercy Clinic Eye Specialists- Ophthalmology, Springfield, Missouri
  - UNMC Truhlsen Eye Institute, Omaha, Nebraska
  - UNC Kittner Eye Center, Chapel Hill, North Carolina
  - Cincinnati Eye Institute, Cincinnati, Ohio
  - OSU Wexner Medical Center, Columbus, Ohio
  - Ophthalmic Partners, PC, Bala-Cynwyd, Pennsylvania
  - Vanderbilt Eye Institute, Nashville, Tennessee
  - Houston Eye Associates, Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - Blanton Eye Institute/Houston Methodist Eye Associates, Houston, Texas
  - Texas Eye Research Center, Hurst, Texas
  - R and R Eye Research, LLC, San Antonio, Texas
  - Piedmont Eye Center, Lynchburg, Virginia
  - WVU Eye Institute, Morgantown, West Virginia
  - The Eye Centers of Racine and Kenosha, Kenosha, Wisconsin
  - University of Wisconsin, Madison, Wisconsin